CLINICAL TRIAL: NCT01101243
Title: How Much UVB Radiation is Necessary to Maintain Summer Vitamin D Level During Winter?
Brief Title: Maintenance of Vitamin D Level by UVB Radiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: The Danish Medical Research Council (Other)
Responsible Party: Morten Bogh MD, Bispebjerg Hospital, Department of Dermatology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H-C-2008-072
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Vitamin D Status
Keywords: Vitamin D; UVB; Frequency; Body surface area; Dose-Response
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Active Comparator): Body surface area: 88 %
  Interventions: Radiation: Broadband UVB
- Group 2 (Active Comparator): Body surface area: 22 %
  Interventions: Radiation: Broadband UVB
- Group 3 (Active Comparator): Body surface area: 88 %
  Interventions: Radiation: Broadband UVB
- Group 4 (Active Comparator): Body surface area: 88 %
  Interventions: Radiation: Broadband UVB
- Group 5 (No Intervention): Body surface area: 0 %
  Interventions: Other: Control group

INTERVENTIONS:
Radiation: Broadband UVB — UVB dose: 1 SED every week
  Arms: Group 1
Radiation: Broadband UVB — UVB dose: 4 SED every second week
  Arms: Group 2
Radiation: Broadband UVB — UVB dose: 1 SED every second week
  Arms: Group 3
Radiation: Broadband UVB — UVB dose: 1 SED every month
  Arms: Group 4
Other: Control group — No intervention
  Arms: Group 5

SUMMARY:
The purpose of the study is to determine the frequency of UVB radiations necessary to maintain the Vitamin D level during winter time.

DETAILED DESCRIPTION:
The work is addressing vitamin D production after UVB exposure and explore how much UVB radiation which is necessary to maintain a sufficient vitamin D level during the winter period in Denmark. 4 different UVB exposure times and 2 different UVB doses to 2 different body surface areas.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* Healthy

Exclusion Criteria:

* Sun bed use
* Holiday or business travel south of 45 degrees latitude during trial
* Illness
* Drug addiction
* Pregnancy
* Lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Vitamin D (nmol/l) | Monthly during 4 months
  Vitamin D measured in a blood sample to define the relationship between frequency of UVB radiations and the Vitamin D level.

SECONDARY OUTCOMES:
Parathyroideahormone (pmol/l) | 4 months
  To investigate whether parathyroideahormone is influenced by the UVB radiations.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Christian Wulf, Professor, Study Chair — Bispebjerg Hospital, Department of Dermatology
Locations (1):
- Bispebjerg Hospital, Copenhagen, NV, Denmark